CLINICAL TRIAL: NCT02453035
Title: X-Pand is Intended to Use the DESolve Scaffold System in Treatment of CAD Patients, by Including "Real World" Use of the DESolve Scaffold Over a Broad Spectrum of Geographies, A Wide Variety of Practicing Clinicians & A Minimum Degree Of Selection Criteria
Brief Title: DESolve® X-Pand Global Post Market Registry
Acronym: X-Pand
Status: Terminated | Type: Observational
Why Stopped: slow enrollment due to change in worldwide scaffold usage
Sponsor: Elixir Medical Corporation (Industry)
Collaborators: European Cardiovascular Research Center (Network)
Responsible Party: Sponsor
Other Study IDs: ELX-CL-1503
Record Dates: First submitted 2015-05-13; First posted 2015-05-25 (Estimated); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Coronary Artery Stenosis
Keywords: bioresorbable scaffold; CAD
MeSH Terms: conditions — Coronary Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PTCA - Desolve Scaffold: Patients with coronary artery stenosis who have been treated with a DESolve bioresorbable coronary scaffold
  Interventions: Device: PTCA - Desolve Scaffold

INTERVENTIONS:
Device: PTCA - Desolve Scaffold — Percutaneous Coronary Artery Intervention with a DESolve bioresorbable coronary scaffold
  Other Names: PTA. PCI

SUMMARY:
The X-Pand Registry is intended to facilitate analysis of acute & long-term safety as well as treatment outcomes with DESolve in patients with CAD.

DETAILED DESCRIPTION:
The Xpand Registry is a single-arm, multi-center, clinical Follow up study of patients with significant coronary stenosis who are treated with a commercially available DESolve Scaffold.

The Registry is an observational study. The patients should be treated according to the current DESolve IFU, professional societies guidelines & internal hospital guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Minimal age 18 years
2. Patient is willing/able to cooperate with study procedures and required follow up visits. Patient or legal representative has been informed & agrees by signing EC approved written consent. Consent can occur before implantation of the DESolve scaffold (planned procedure) or within 30 days post implantation procedure for retrospective enrollment (unplanned procedure).
3. Planned or unplanned DESolve scaffold implantation

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who have received implants of one or more DESolve scaffold(s)
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2015-05-13 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
TLF (Target Lesion Failure) | 12 months
  TLF is defined as: cardiac death, MI not clearly attributable to a non-intervention vessel, and clinically-indicated target lesion revascularization (TLR)
Death | 12 months
  All cause mortality
MI | 12 months
  Myocardial Infarction
CABG | 12 months
  Emergency bypass surgery (CABG)
CD-TVR | 12 months
  Clinically-driven revascularization of the target vessel (Target Vessel Revascularization, TVR) using percutaneous or surgical methods (CABG)

SECONDARY OUTCOMES:
Thrombosis | 12 months
  Thrombosis: The ARC stent thrombosis criteria are applied
Device Success | day of treatment procedure
  Successful delivery and deployment of the Clinical Investigation scaffold at the target lesion and successful withdrawal of the scaffold delivery system with attainment of final residual stenosis < 50% by QCA (by visual estimation if QCA is unavailable). Standard pre-dilation catheters and post-dilatation catheters (if applicable) may be used. Bailout subjects will be included as device success only if the above criteria for clinical device success are met
Procedure Success | 30 days
  Successful delivery and deployment of the DESolve scaffold at the target lesion and successful withdrawal of the scaffold delivery system with attainment of final residual stenosis of < 50% by QCA (by visual estimation if QCA unavailable) and/or using any adjunctive device without the occurrence of ischemia driven major adverse cardiac event (MACE) during the hospital stay with a maximum of first seven days post index procedure.
MACE | 3 years
  MACE is defined as: cardiac death, MI not clearly attributable to a non-intervention vessel, and clinically-indicated target lesion revascularization (TLR)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Fajadet, Dr., Principal Investigator — University Hospital of Toulouse; Holger Nef, Prof Dr., Principal Investigator — Universitätsklinikum Giessen und Marburg
Locations (5):
- Germany (4):
  - Kerckhoff-Klinik, Bad Nauheim
  - Universitätsklinikum Giessen, Giessen
  - GPR Klinikum Rüsselsheim, Rüsselsheim am Main
  - Krankenhaus der Barmherzigen Brüder, Trier
- St. Antonius Ziekenhuis, Nieuwegein, Netherlands